CLINICAL TRIAL: NCT06432998
Title: Oncological Perineal Massage in Vaginal Stenosis and Dyspareunia in Women With Gynecological Cancer
Brief Title: Perineal Massage in Women With Gynecological Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUNSC_2023_104
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Cancer Pain; Neck Cancer
MeSH Terms: conditions — Cancer Pain; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perineal massage (Experimental): Ten sessions of perineal massage, which will be carried out for fifty minutes, once a week, together with a health education program.
  Interventions: Other: Perineal massage
- Treatment with dilators (Active Comparator): A health education session will be held but then the use of vaginal dilators will be done according to the gold standard treatment.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Perineal massage — The technique will be applied for approximately twenty minutes and will be carried out as follows: the vaginal dilator is introduced progressively using crescent-shaped movements. Once the dilator is fully inserted, movements will be made from bottom to top and from one side to the other, and then continue with the crescent-shaped movements.
  Arms: Perineal massage
Other: Standard treatment — The treatment will consist of the use of vaginal dilators according to the gold standard proposed in the literature. It will consist of introducing the same dilators as for the experimental group, with the same time schedule, but without massage, only introducing the dilator and keeping it in the vagina for 20 minutes.
  Arms: Treatment with dilators

SUMMARY:
The high incidence of gynecological cancers, together with dyspareunia and vaginal stenosis, some of its most frequent sequelae, create the need to continue studying and researching oncological physiotherapy techniques that treat and prevent these sequelae, in order to preserve and/or improve the quality of life of cancer patients. Therefore, through this study, we sought to verify the effectiveness of oncological perineal massage to treat pain during sexual intercourse and vaginal stenosis.

The objective of this study will be to demonstrate the effectiveness of a treatment that will consist of a health education session related to the pelvic floor and the consequences related to cancer along with ten sessions of oncological perineal massage that will be carried out for fifty minutes, once a week.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 52 years old
* Oncology patients with a diagnosis of dyspareunia and vaginal stenosis related to treatments.
* Patients with QT/RT/BT treatment who have a diagnosis of dyspareunia and vaginal stenosis.
* Patients on hormonal suppressive treatment with a diagnosis of dyspareunia and vaginal stenosis.

Exclusion Criteria:

* Patients who do not accept intracavitary treatment.
* Patients with abdominopelvic surgical treatment prior to oncological process.
* Patients with a diagnosis of dyspareunia prior to cancer.
* Patients with vaginal narrowing prior to cancer.
* Patients with menopause at the time of cancer diagnosis

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women diagnosed with vaginal stenosis and dyspareunia due to cancer
Enrollment: 35 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Pain (Visual Analoge Scale) | Change from baseline at six months
  Visual Analogical Scale (VAS) is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured orientated from the left "0" (worst) to the right "10"(best)

SECONDARY OUTCOMES:
Criteria for Adverse Events (CTCAE) | Change from baseline at six months
  Grade refers to the severity of the Adverse Events. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on a general guideline where grade 1 and grade 5 are the best and worst result respectively.
Quality of life (EORCT QLQ-C30) | Change from baseline at six months
  The EORTC QLG Core Questionnaire (EORTC QLQ-C30) is a 30-item instrument designed to measure quality of life in all cancer patients. The scores obtained can have values between 0 and 100, which determines the level of impact of the cancer on the patient of each of the scales. High values on the global health and function status scales indicate a better quality of life, while on the symptoms scale it would indicate a decrease in quality of life since it indicates the presence of symptoms associated with cancer.
Female sexual function index | Change from baseline at six months
  Female sexual function index (FSFI) is a survey measuring the sexual functioning of women in six different domains: desire, arousal, lubrication, orgasm, satisfaction and pain.The items are then scaled to achieve a maximum score of 36.
Likert questionnaire by sexual dysfunction | Change from baseline at six months
  Likert scales are a structured way for researchers to gather diverse opinions and attitudes. They allow respondents to express agreement, disagreement, or neutrality concerning statements or questions. The scale values range from 1 to 5, with 1 being the worst result and 5 being the best result.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Perez-García, Principal Investigator — Asociación Española Contra el Cáncer en la provincia de Santa cruz de Tenerife.
Locations (1):
- Asociación Española Contra el Cáncer en la provincia de Santa cruz de Tenerife., Santa Cruz de Tenerife, Tenerife, Spain

REFERENCES:
- [Derived] Perez-Garcia R, Abuin-Porras V, Minguez-Esteban I, Pecos-Martin D. Oncological perineal massage in vaginal stenosis and dyspareunia in women with gynecological cancer: a randomized controlled trial. Front Oncol. 2025 Nov 28;15:1680126. doi: 10.3389/fonc.2025.1680126. eCollection 2025. PMID 41395600